CLINICAL TRIAL: NCT03381261
Title: Novel Concepts for OnabotulinumtoxinA (Botox) Mechanisms of Action: Role in Altering the Molecular Environment in Which Pain Fibers Exist
Brief Title: (Botox) Mechanisms of Action in Altering the Molecular Environment in Which Pain Fibers Exist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, William Gerald Austen, Chief, Plastic and Reconstructive Surgery; Chief, Burn Surgery, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2017P001813
Record Dates: First submitted 2017-12-18; First posted 2017-12-21 (Actual); Results first posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Migraine
Keywords: chronic migraine; trigeminal neuralgia; migraine surgery; nerve decompression
MeSH Terms: conditions — Migraine Disorders; Trigeminal Neuralgia | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Botulinum toxin type A injection arm (Experimental): All patients will be injected with Botulinum toxin on one side of the back of the head.
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Injection of Botulinum toxin type A in back of head
  Other Names: Botox

SUMMARY:
To compare Botox-treated and Botox-untreated symptomatic tissues (defined as areas where the head hurts and the pain is felt) of chronic migraine (CM) patients using molecular studies.

DETAILED DESCRIPTION:
Eligible patients for migraine surgery will be injected unilaterally with Botox prior to surgery. The effects of Botox on tissues will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Diagnosis of Chronic Migraine consistent with International Classification of Headache Disorders (ICHD-III) criteria, with a history of bilateral headache pain and chronic tenderness in neck muscles
* Patient is capable and willing to provide informed consent
* Female subjects of child bearing potential must have a negative pregnancy test at enrollment and agree to remain abstinent or use acceptable methods of birth control (i.e., hormonal contraceptives, inrauterine device, diaphragm with spermicide, cervical cap or sponge, condoms or partner has had a vasectomy) for three months following injections of Botox
* Patients referred by their primary Neurologist to the study surgeon and who are determined to be candidates for surgical decompression of extracranial sensory nerves.
* Patient agrees to abstain from protocol-specific excluded medications beginning 14 days prior to the decompression surgery.

Exclusion Criteria:

* Patient has hypersensitivity reactions or other intolerance to Botox
* Patient is pregnant or trying to become pregnant with the timeframe of the study.
* Infection at proposed injection sites.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William G. Austen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: One side on the occipital head
Groups:
- Treatment With Onabotulinumtoxin A Injection: One side of the occipital head of participants was treated with a total of 40 units of onabotulinumtoxin A injection 30 days prior to their scheduled, study-unrelated, nerve decompression surgery.
  The specific sites injected were the following:
  * 2 sites in the Occipitalis muscle (5 units each)
  * 4 sites in the Cervical Paraspinal muscle group (5 units each)
  * 2 sites in the Trapezius muscle (5 units each)
  The selection of the side of the head to receive the injection treatment was random based on subject number. Participants assigned odd numbers were injected on the right, while participants with even numbers were injected on the left side.
- No Treatment: The other side of the occipital head of participants did not receive any injection intervention.
Period: Pre-Transcriptomic Analysis
Arm/Group | Treatment With Onabotulinumtoxin A Injection | No Treatment
Started | 37; 37 One side on the occipital head (In this split-person study, a total of 37 participants were enrolled and started the study. For each patient, two sides of the head were each assigned to a different intervention. The unit of measure for the study was "side of head".) | 37; 37 One side on the occipital head (In this split-person study, a total of 37 participants were enrolled and started the study. For each patient, two sides of the head were each assigned to a different intervention. The unit of measure for the study was "side of head".)
Split-Person Intervention (The split-person intervention consisted in injecting onabotulinumtoxinA in one side of the occipital head and no injection treatment on the other side.) | 32; 32 One side on the occipital head (Among the 37 participants who were enrolled, consented and started the study, 32 patients underwent the split-person intervention which consisted in injecting onabotulinumtoxinA in one side of their head and no injection treatment on the other side.) | 32; 32 One side on the occipital head (Among the 37 participants who were enrolled, consented and started the study, 32 patients underwent the split-person intervention which consisted in injecting onabotulinumtoxinA in one side of their head and no injection treatment on the other side.)
Migraine Surgery (Participants underwent nerve decompression migraine surgery 30 days following the split-person intervention. During surgery, discarded tissue was collected for transcriptomic analyses.) | 31; 31 One side on the occipital head (Among the 32 patients who underwent the split-person intervention, 31 underwent nerve decompression migraine surgery within 30 days. Thus, tissue from both sides of the head was collected for 31 patients.) | 31; 31 One side on the occipital head (Among the 32 patients who underwent the split-person intervention, 31 underwent nerve decompression migraine surgery within 30 days. Thus, tissue from both sides of the head was collected for 31 patients.)
Completed | 31; 31 One side on the occipital head (A total of 31 participants completed the study (screened, consented, underwent onabotulinumtoxinA injection on one side of the head and no injection on the other side, underwent nerve decompression surgery, had tissues collected from both sides of occipital head).) | 31; 31 One side on the occipital head (A total of 31 participants completed the study (screened, consented, underwent onabotulinumtoxinA injection on one side of the head and no injection on the other side, underwent nerve decompression surgery, had tissues collected from both sides of occipital head).)
Not Completed | 6; 6 One side on the occipital head | 6; 6 One side on the occipital head
Period: Transcriptomic Analysis
Arm/Group | Treatment With Onabotulinumtoxin A Injection | No Treatment
Started | 31; 31 One side on the occipital head | 31; 31 One side on the occipital head
Completed | 18; 18 One side on the occipital head (Among the 31 patients who had tissues collected from both sides of their heads, 18 patients had tissues that were collected which fulfilled all criteria for inclusion for transcriptome analyses and data interpretation following transcriptomic data quality, background thresholding and normalization zesting. The 13 patients who were not included in the analysis are those whose transcriptome data quality failed inclusion criteria.) | 18; 18 One side on the occipital head (Among the 31 patients who had tissues collected from both sides of their heads, 18 patients had tissues that were collected which fulfilled all criteria for inclusion for transcriptome analyses and data interpretation following transcriptomic data quality, background thresholding and normalization zesting. The 13 patients who were not included in the analysis are those whose transcriptome data quality failed inclusion criteria.)
Not Completed | 13; 13 One side on the occipital head | 13; 13 One side on the occipital head

BASELINE CHARACTERISTICS:
Population: In this split-person study, a total of 18 patients were analyzed. The unit of measure was each side of the head which were assigned to treatment arm or no treatment arm.
  Among 37 total participants enrolled, 31 received the split-person treatment, underwent surgery and had tissues collected. Tissues of 18 patients fulfilled all criteria for inclusion for transcriptome analyses and data interpretation (data quality, background thresholding and normalization).
Units Other Than Participants: Sides of head
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment With Onabotulinumtoxin A Injection | No Treatment | Total
Number analyzed (Participants) | 18 | 18 | 18
Number analyzed (Sides of head) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants] — The average age of the patient population was 45 years old (standard deviation 14 years). Patient age range was 21 to 74 years old. Population: Among 37 total participants enrolled, 31 received the split-person intervention, underwent surgery, and had tissues collected from both sides. Among the 31, tissues of 18 patients fulfilled all criteria for inclusion for transcriptome analyses and data interpretation (data quality, background thresholding and normalization). Therefore, a total of 18 participants were included in the analysis.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 17 | 17 | 34
    >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (14) | 45 (14) | 45 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 17 | 34
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: Participants]
  United States | 18 | 18 | 18
Monthly migraine days [Mean (Standard Deviation); unit: days per month] | 19 (10) | 19 (10) | 19 (10)

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Gene Expression in Chronic Migraine Patients With OnabotulinumtoxinA Injection Treatment Versus No Treatment
Description: In this split-person study, patients with chronic bilateral occipital migraines scheduled for a study-unrelated migraine surgery (occipital nerve decompression surgery) had one side of their head undergo treatment with onabotulinumtoxinA injection, while the other side of the head underwent no treatment. Occipital periosteum tissue of both injected and uninjected sides was collected during migraine surgery for targeted transcriptome profiling and genome-wide epigenome analyses of inflammatory gene expression using NanoString of 594 genes (579 immunology-related genes involved in adaptive/innate response, lymphocyte activation, cytokine/chemokine/NF-kB/TNF/interferon signalling, neutrophils, macrophages, cytotoxic T, NK, Th1, B and dendritic cells, and 15 internal reference controls). The effects size (ratio of geometric means) of expression of gene expression was evaluated between injected and uninjected sides.
Time Frame: One year
Population: Among 37 total participants enrolled, 31 completed the study (received botox injection on one side, underwent surgery, had tissues collected from both sides). Among the 31, tissues of 18 patients fulfilled all criteria for inclusion for transcriptome analyses and data interpretation (data quality, background thresholding and normalization). The 13 patients who completed the study but were not included in the analysis are those whose transcriptome data quality failed inclusion criteria.
Measure: Median (Inter-Quartile Range); unit: mRNA units
Units Other Than Participants: Sides of head
Groups:
- Treatment With OnabotulinumtoxinA Injection: One side of the occipital head of participants was treated with a total of 40 units of onabotulinumtoxinA injection 30 days prior to their scheduled, study-unrelated, nerve decompression migraine surgery.
  The specific sites injected were the following:
  * 2 sites in the Occipitalis muscle (5 units each)
  * 4 sites in the Cervical Paraspinal muscle group (5 units each)
  * 2 sites in the Trapezius muscle (5 units each)
  The selection of the side of the head to receive the injection treatment was random based on subject number. Participants assigned odd numbers were injected on the right, while participants with even numbers were injected on the left side.
Arm/Group | Treatment With OnabotulinumtoxinA Injection | No Treatment
Number analyzed (Participants) | 18 | 18
Number analyzed (Sides of head) | 18 | 18
mRNA units | 44.46156 [12.98994 to 137.8325] | 68.74241 [26.35755 to 191.9613]
Statistical Analysis 1: Comparison: Treatment With OnabotulinumtoxinA Injection vs No Treatment; Test type: Other — While descriptive statistics were presented in the original mRNA units using median and interquartile range (25th, 75th), statistical group comparison and effect sizes were reported as the ratio of the geometric means; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: For each patient, from the time of informed consent to 6 years following surgery, self-reported adverse events were reviewed by the study physician during patient contact and follow-ups.
Arm/Group | Botulinum Toxin Type A Injection Arm
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT03381261/Prot_SAP_000.pdf